CLINICAL TRIAL: NCT00291850
Title: Phase II Trial of Dose-dense Paclitaxel and Cisplatin as Neo-adjuvant Chemotherapy for Operable Stage II and IIA Non-Small Cell Lung Cancer
Brief Title: Phase II Trial of Dose-dense Paclitaxel and Cisplatin as Neo-adjuvant Chemotherapy for Operable Stage II and IIA NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: no patient recruitment
Sponsor: Central European Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CECOG/NSCLC.3.2.002
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Cisplatin; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Paclitaxel, Cisplatin, Pegfilgrastim

SUMMARY:
A single arm, open-label phase II is appropriate to evaluate the efficacy and safety of dose - dense combination of paclitaxel with cisplatin supported by pegfilgrastim for neo-adjuvant chemotherapy in this patient population.

DETAILED DESCRIPTION:
This is an open-label, single-arm Phase II study of dose-dense regimen with paclitaxel and cisplatin supported by pegfilgrastim as neo-adjuvant chemotherapy in patients with operable stage II, IIA NSCLC.

Paclitaxel will be administered via intravenous infusion over approximately 3 hours at dose of 175mg/m2 on Day 1 of each 14-day cycle. Cisplatin 75mg/m2 will be given via intravenous infusion on day 1 (after paclitaxel) according to institutional guidelines.

Pegfilgrastim (Neulasta) fixed dose of 6mg (0.6mL of a 10mg/mL solution) as a single subcutaneous injection on Day 2 of each study cycle.

All drugs will be given in 2-weekly cycle. Three cycles of pre-operative chemotherapy are planned.

ELIGIBILITY:
Inclusion Criteria:

* histologic or cytologic diagnosis of NSCLC
* Presence of clinical Stage IIA,IIB or IIA disease
* tumor amenable to curative surgical resection
* Patients with clinically measurable lesions will be enrolled in this study.
* No prior tumor therapy
* Performance status of 0-1 on ECOG Scale
* Patients compliance and geographic proximity that allow adequate follow-up.
* Medical fitness of patient, including respiratory function, adequate for radical NSCLC surgery.

Exclusion Criteria:

* Presence of clinical Stage IIIA disease, according to the revision by Mountain CF of American Joint Committee on Cancer.
* Treatment within the last 30 days with any investigational drug.
* Cocurrent administration of any other tumor therapy, including radiotherapy, cytotoxic chemotherapy, immunotherapy, molecular target therapy.
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* pregnancy/breast feeding
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patients ability to complete the study, at the discretion of the investigator.
* poorly controlled diabetes mellitus
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* History of significant neurological or mental disorder, including seizures or dementia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-06

PRIMARY OUTCOMES:
the evaluation of the clinical response rate of neo-adjuvant chemotherapy with dose-dense therapy of paclitaxel and cisplatin(PC) with peg-filgrastim in patients with operable NSCLC

SECONDARY OUTCOMES:
>To evaluate the safety of neo-adjuvant chemotherapy with PC
- to characterize the toxicity of PC, include febrile neutropenia.
- to evaluate peri- and post-operative mortality
> to determine the pathological complete response rate
> to determine the complete tumor resection rate
> to evaluate proportion of cycle 2 and all cycles chemotherapy given with planned dose-on-time and proportion of patients receiving planned dose-on-time in cycle 2 and over all cycles.
> To evaluate the following time-to-event efficacy variables:
- disease free survival
- overall survival
> to evaluate Quality of life (EORTC QLQ-C30 and QLQ-LC13)

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Krzakowski, MD, Principal Investigator — M.Sklodowska-Curie Memorial, Dep of Lung and Thoracic Tumours, Warsaw
Locations (5):
- AKH, Universitätsklinik für Innere Medizin 1, Vienna, Austria
- Hungary (2):
  - Somogy Country Pulmo and Cardio Hospital,, Mosdós
  - Markusovszky Hospital, Szombathely
- Poland (2):
  - M. Sklodowska-Curie Memorial Dep. Of Lung and Thoracic Tumours,, Warsaw
  - Klinika Chirurgii Instytutu Gruzlicy i Chorob Pluc, Warsaw